CLINICAL TRIAL: NCT05802251
Title: Sonographic Parameters and Risk of Antepartum Hemorrhage in Asymptomatic Women With Placenta Previa: A Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maya Abdelrazek, Lecturer, Ain Shams University
Other Study IDs: MD 172 2022
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonographic parameters — cervical length. placental thickness. distance placental edge from internal os of the cervix

SUMMARY:
The aim of this study is to evaluate the effectiveness of ultrasonographic parameters (cervical length, placental thickness and distance placental edge from internal os of the cervix) in predicting the risk of antepartum hemorrhage and emergency cesarean delivery in asymptomatic women with placenta previa.

DETAILED DESCRIPTION:
The incidence of placenta previa is 3-5 per 1000 pregnancies worldwide and is still rising because of increased maternal age, parity, cesarean section rates, assisted reproductive technology, maternal smoking with the widespread use of transvaginal ultrasound. antepartum hemorrhage is an important cause of maternal and neonatal morbidity and mortality in pregnant women with placenta previa. However, the epidemiological characteristics are not completely understood. this study aims at evaluating the sonographic findings in asymptomatic women with placenta previa as cervical length, placenta thickness and distance from cervix to placental edge to recommend management for in-patients versus out-patient antenatal care and early planned hospital admission and delivery for women at high risk of antepartum hemorrhage and preterm cesarean section and hysterectomy for life threatening antepartum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic women diagnosed with placenta previa according to RCOG (GTG No. 27a, 2018): placenta lies directly over the internal os for pregnancies more than 16 weeks' gestation on transabdominal or transvaginal scanning.
* Gestational age between 28 till 37 weeks' gestation (as delivery should be considered between 36 and 37 weeks of gestation for women presenting with uncomplicated placenta previa)

Exclusion Criteria:

* Multiple pregnancies.
* Threatened preterm labor or preterm rupture of membranes.
* History of bleeding in the current pregnancy.
* Polyhydraminos (AFI > 25 cm).
* History of cervical surgery (cone biopsy).
* Presence of cervical cerclage.
* Maternal use of vaginla progesterone.
* History of maternal disease (hypertensive, DM, Cardiac).
* Fetal malformation or growth restriction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Asymptomatic pregnant women diagnosed with placenta previa between 28 to 37 weeks' gestation.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
maternal bleeding rate | till delivery
  number of attacks of antepartum hemorrhage

SECONDARY OUTCOMES:
Blood transfusion | till delivery 36 to 37 weeks
  number of PRBCs
Emergency Cesarean section | till delivery 36 to 37 weeks
  severe antepartum hemorrhage requiring delivery
Premature delivery | 37 week's gestation
  before the planned delivery date (before 37 weeks' gestation)
Need for cesarean hysterectomy | during cesarean section
  cesarean hysterectomy due to bleeding or placenta accreta spectrum
Postpartum hemorrhage | Within 2 hours of delivery
  severity of attacks and required further management or blood transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt